CLINICAL TRIAL: NCT06556641
Title: Phase Ib Clinical Study on the Safety, Tolerance, Pharmacokinetics, and Pharmacodynamics of GZR33 and GZR101 in Healthy Adult Male Subjects
Brief Title: A Clinical Study of GZR33 and GZR101 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GZR-CH1013
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Part A : randomized, open-label, single-dose, two-sequence, two-period, cross-over
  Single administration of GZR33, washout period of 14 days, followed by single administration of Insulin Degludec
  Single administration of Insulin Degludec, washout period of 14 days, followed by single administration of GZR33
  Interventions: Drug: GZR33 Injection; Drug: Insulin Degludec
- Part B (Experimental): Part B: randomized, double-blind, placebo-controlled, multiple-dose, parallel
  Drug: GZR33 Injection Participants will receive once daily GZR33 Injection or placebo for 6 days, s.c.
  Drug: GZR101 Injection Participants will receive once daily GZR101 Injection or placebo for 6 days, s.c.
  Interventions: Drug: GZR33 Injection; Drug: GZR101 Injection; Drug: Placebo

INTERVENTIONS:
Drug: GZR33 Injection — Administered as once daily subcutaneous dose
Drug: GZR101 Injection — Administered as once daily subcutaneous dose
  Arms: Part B
Drug: Placebo — Administered as once daily subcutaneous dose
  Arms: Part B
Drug: Insulin Degludec — Administered as once daily subcutaneous dose
  Arms: Part A

SUMMARY:
This study evaluates the safety, tolerability, pharmacokinetics, and pharmacodynamics of GZR33 and GZR101 in healthy adult male subjects.This study consists of Part A and Part B.

Part A is a randomized, open-label, single-dose, two-sequence, two-period, cross-over design comparative study evaluating the PD and PK characteristics of GZR33 and Insulin Degludec Injection.

Part B is a randomized, double-blind, placebo-controlled, multiple-dose, parallel-group design study evaluating the safety, tolerability, immunogenicity, and PK of GZR33 and GZR101.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participated in the study and signed the informed consent form (ICF);
* 2.Chinese healthy male adult subjects aged 18-45 years old (including 18 and 45 years old as of the date of signing the ICF);
* 3.During screening period, the body mass index (BMI) between 19.0 and 24.0 kg/m2, inclusive, and a body weight>50 kg (not containing 50kg).

Exclusion Criteria:

* 1.History of drug abuse within one year prior to screening.
* 2.History of alcohol abuse within 6 months prior to screening (alcohol abuse is defined as more than 14 units weekly: 1 unit of alcohol equals to 360 mL of beer, 150 mL of wine, or 45 mL of 40% alcohol).The subject who smoke more than 5 cigarettes per day within 3 months prior to screening, smoke within 48 h prior to the use of the investigational drug, and is unwilling to refrain from smoking and drinking during the trial period.
* 3.Allergic constitution, or history of bronchial asthma, hives, eczema and other allergic diseases (except mild asymptomatic seasonal allergy), or known allergy to the investigational drug or its excipients, hypersensitivity or intolerance.
* 4.Hepatitis B surface antigen (HBsAg), hepatitis C antibodies, syphilis spiral test or human immunodeficiency virus (HIV) antibodies positive.
* 5.History of needle and blood sickness, and subject couldn't tolerate venipuncture for blood collection, or be difficult to collect blood.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-12-17 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
AUC0-24h | From 0 to 24 hours
  Area under the plasma concentration-time curve from time 0 to 24 hours
Incidence of adverse events (AE) | From Predose to Day12
  Any changes or abnormal results in the following safety variables: incidence of adverse events (AE), including but not limited to hypoglycemic reactions, injection site reactions, clinical laboratory tests, 12-lead ECG, vital signs, physical examination, and local tolerability at the injection site.

SECONDARY OUTCOMES:
Cmax | From Predose to Day7
  Maximum plasma concentration
tmax | From Predose to Day7
  Time to reach maximum plasma concentration
AUC0-last | From Predose to Day7
  Area under the plasma concentration-time curve from time 0 to the last blood sampling time point

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Study Site, Xingtai, Hebei, China

IPD SHARING:
Plan to Share IPD: No